CLINICAL TRIAL: NCT03192124
Title: Evaluating Bactisure Wound Lavage in Cleansing Orthopedic Surgical Wounds
Brief Title: Evaluating Bactisure Wound Lavage in Orthopedic Wounds
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: H.CR.I.AM.16.10
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Infection of Total Knee Joint Prosthesis
Keywords: primary total knee; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Level 1 Panel is a quantitative real-time PCR test to detect 12 microbial organisms that may be present in patient specimen (bacteria and fungi) and includes test for resistance factors to vancomycin and methicillin.
  Microbial DNA in each sample will be sequenced using the Ion Torrent PGM sequencer in order to establish what type of bacterial and fungal species are present.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Bactisure — Level 1 Panel is a quantitative real-time PCR test to detect 12 microbial organisms that may be present in patient specimen (bacteria and fungi) and includes test for resistance factors to vancomycin and methicillin.
  Microbial DNA in each sample will be sequenced using the Ion Torrent PGM sequencer in order to establish what type of bacterial and fungal species are present.

SUMMARY:
To demonstrate a reduction of debris in knee synovial fluid as demonstrated by WBC cell counts before and after irrigation with Bactisure Wound Lavage.

DETAILED DESCRIPTION:
This study will demonstrate a reduction in fluid cell counts in aspirate acquired from primary total knee arthroplasty patients diagnosed with infection. WBC cell counts will be compared before and after articular irrigation with Bactisure Wound Lavage.

This study is a prospective, multi-center, single arm study involving orthopedic surgeons skilled and experienced in deep surgical debridement and in I & D or reoperation (revision) total knee arthroplasty procedures. A maximum of seven study centers will enroll a maximum of 40 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing I & D or reoperation (revision) surgery for an infected primary TKA.
* Patient is 18 years of age or greater.
* Patient is skeletally mature.
* Occurs within 30 days of the operation or within 1 year or more if an implant is present
* Involves deep soft tissues (e.g., fascia and/or muscle) of the incision
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the protocol

Exclusion Criteria:

Patients will be excluded from this study if:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Known sensitivity or allergic reaction to benzalkonium chloride one or more of the solvent, chelating agent, or buffer in the solution
* Multiple (>1) infected implants
* Medically unfit for irrigation & debridement procedure
* Pregnancy
* The patient is:
* prisoner
* mentally incompetent or unable to understand what participation in the study entails
* anticipated to be non-compliant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential Subjects (M and F, age 18 years or older) diagnosed with Prosthetic Joint Infection (PJI) following primary total knee (TKA) implantation, who are undergoing I & D or reoperation (revision) surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Reduction WBC | Intraoperative
  To demonstrate a reduction of debris in knee synovial fluid as demonstrated by WBC cell counts before and after irrigation with Bactisure Wound Lavage

SECONDARY OUTCOMES:
Bacteria Identification | One Week
  To quantitatively and qualitatively assess the synovial fluid for the presence of bacteria prior to and after lavage. This testing will compare the microbial population (species) of the surgical wounds by serial culture dilution, and bacterial identification by PCR before and after irrigation.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, MBA, Study Director — Zimmer Biomet
Locations (5):
- United States (5):
  - LA Orthopedic Institute, Los Angeles, California
  - University of Kentucky Orthopedic Spine & Total Joint Service, Lexington, Kentucky
  - Norton Orthopaedic & Sports Medicine Specialists, Louisville, Kentucky
  - The Cleveland Clinic, Cleveland, Ohio
  - The Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No